CLINICAL TRIAL: NCT04085718
Title: Evaluation of the feaSibility of FDG-PET/CT Images Comparing to MRI and Endomyocardial Biopsy Findings in clinicAlly Suspected Myocarditis
Brief Title: FDG-PET/CT Images Comparing to MRI and Endomyocardial Biopsy in Myocarditis
Acronym: STREAM
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Krzysztof Ozieranski, Principal Investigator, Medical University of Warsaw
Other Study IDs: STREAM
Record Dates: First submitted 2019-09-08; First posted 2019-09-11 (Actual); Last update posted 2019-09-13 (Actual); Status verified 2019-09

CONDITIONS: Myocarditis
Keywords: endomyocardial biopsy; myocarditis; anti-heart autoantibodies; biomarker; positron emission computed tomography; heart failure; cardiomyopathy; magnetic resonance imaging
MeSH Terms: conditions — Myocarditis; Heart Failure; Cardiomyopathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum stored at -80 degrees celsius
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study arm: All included patients will undergo FDGPET/CT scan

SUMMARY:
Fifty hospitalized consecutive patients with clinically suspected myocarditis (MC) who meet the inclusion/exclusion criteria will be enrolled to the study.

During index hospitalization patients will undergo a standard clinical evaluation (physical examination, collection of a medical history, blood tests (including troponin, N-terminal-pro Brain Natriuretic Peptide (NTproBNP), C-reactive protein (CRP), Suppression of Tumorigenicity 2 (ST2), Galectin-3), 24-h Holter ECG, echo, coronary angiography, magnetic resonance imaging (MRI)). Women of childbearing potential will undergo a pregnancy test prior to radiological examinations. After signing the informed consent patients will undergo resting single photon emission computed tomography (SPECT) to assess possible myocardial perfusion defects and then 18F-2-fluoro-2-deoxy-D-glucose fluorodeoxyglucose positron emission tomography/computed tomography FDG-PET/CT. After MRI and FDG-PET/CT tests patients will undergo right ventricular endomyocardial biopsy (EMB) (5-8 myocardial tissue samples). Blood biomarkers of fibrosis and myocardial necrosis, as well as anticardiac autoantibodies will be evaluated at baseline and after 3 months (serum will be stored at -80 °C for final evaluation). After 3-months from enrollment follow-up visit will be performed with clinical evaluation. All patients will undergo physical examination, collection of a medical history, blood tests, 24-h Holter ECG, echo, MRI.

DETAILED DESCRIPTION:
Fifty hospitalized consecutive patients with clinically suspected MC who meet the inclusion/exclusion criteria will be enrolled to the study.

During index hospitalization patients will undergo a standard clinical evaluation (physical examination, collection of a medical history, blood tests (including troponin, N-terminal-pro Brain Natriuretic Peptide (NTproBNP), C-reactive protein (CRP), Suppression of Tumorigenicity 2 (ST2), Galectin-3), 24-h Holter ECG, echo, coronary angiography, MRI). Women of childbearing potential will undergo a pregnancy test prior to radiological examinations. After signing the informed consent patients will undergo resting single photon emission computed tomography (SPECT) to assess possible myocardial perfusion defects and then cardiac FDG-PET/CT. After MRI and FDG-PET/CT tests patients will undergo right ventricular EMB (5-8 myocardial tissue samples). Blood biomarkers of fibrosis and myocardial necrosis, as well as anti-heart autoantibodies will be evaluated at baseline and after 3 months (serum will be stored at -80 °C for final evaluation). After 3-months from enrollment follow-up visit will be performed with clinical evaluation. All patients will undergo physical examination, collection of a medical history, blood tests, 24-h Holter ECG, echo, MRI.

FDG-PET/CT imaging Resting SPECT will be performed one day before the FDG-PET/CT examination. Physiological glucose uptake in the myocardium will be suppressed using dietary preparation (low-carbohydrate high-fatty diet). 48 h before the FDG-PET/CT examination, all patients' meals will be low-carbohydrate. 24 h before the FDG-PET/CT examination (the "SPECT day"), breakfast and dinner (last meal at 4:00 PM) will be high-fat, then fasting (a patient should drink only still water) until FDG-PET/CT examination in the next morning (9:00 PM). Single-dose heparin will be administered intravenously at a low dose (50 IU/kg) 15 minutes before the start of the FDG-PET/CT examination to increase the accuracy of the test. Capillary blood glucose level will be measured 20 minutes before the FDG-PET/CT examination.

Because of radiation, for about 6 h after the scan patients should avoid contact with children and pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent (including consent for MRI, FDG-PET/CT and EMB)
* Age ≥18 years
* Clinically suspected MC (according to the 2013 Criteria of the ESC Working Group on Myocardial and Pericardial Diseases)
* Symptoms associated with MC with a duration of <6 months
* Women of childbearing potential must have a negative urine or blood pregnancy test

Exclusion Criteria:

* Pregnancy or lactation
* Any contraindication or intolerance to MRI or PET investigations (including but not limited to: presence of pacemakers not compatible with MRI, aneurysm clips, artificial heart valves, ear implants, or foreign metal objects in the eyes, skin, or body that would contraindicate an MRI scan)
* Subjects with body mass index >45 kg/m2
* Active neoplasm or diagnosed sarcoidosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 50 patients with suspected myocarditis
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-09 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of FDG-PET/CT imaging in diagnosis of MC | baseline
  assessment of sensitivity and specificity of FDG-PET/CT imaging in diagnosis of MC with baseline MRI as a reference

SECONDARY OUTCOMES:
Number of adverse events in the study group. | 3 months
  Association of FDG-PET/CT images with occurrence of heart failure, heart failure hospitalizations, heart failure outpatients visits, MC recurrence, heart transplantation, ventricular or supraventricular arrhythmias.
Correlation of FDG-PET/CT images with EMB results. | baseline
  Correlation of FDG-PET/CT images with EMB results (presence of myocardial inflammation, fibrosis) in patients with clinical suspicion of MC.
Correlation of FDG-PET/CT images with MRI and echo results. | baseline
  Correlation of FDG-PET/CT images with MRI (EGE, LGE, edema) and echo (scar, function left and right ventricles) results assessed at baseline.
Correlation of FDG-PET/CT images with MRI and echo results. | 3 months
  Correlation of FDG-PET/CT images with MRI (EGE, LGE, edema) and echo (scar, function left and right ventricles) results assessed after 3 months.
Correlation of FDG-PET/CT images with the concentration of biomarkers of fibrosis and myocardial necrosis. | 3 months
  Correlation of FDG-PET/CT images with the concentration of biomarkers of fibrosis and myocardial necrosis (troponin, N-terminal-pro Brain Natriuretic Peptide (NTproBNP), C-reactive protein (CRP), Suppression of Tumorigenicity 2 (ST2), Galectin-3) evaluated at baseline and after 3 months.
Correlation of FDG-PET/CT images with the presence and concentration of anti-heart autoantibodies. | 3 months
  Correlation of FDG-PET/CT images with the presence and concentration of anti-heart autoantibodies evaluated at baseline and after 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Marcin D Grabowski, Professor, Study Chair — Medical University of Warsaw

IPD SHARING:
Plan to Share IPD: Yes
External requests for study data will be granted, however, any information that is shared will be blinded to any identifying participant information.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: after end of the study
Access Criteria: External requests accepted by the study investigators